CLINICAL TRIAL: NCT00891488
Title: Systemic and Localized Stress Resilience in Aging: Effects of Physical Fitness
Brief Title: Stress Resilience Study
Status: Completed | Type: Observational
Sponsor: Kronos Longevity Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Tinna Traustadóttir, Ph.D., Associate Director, Exercise Sciences, Kronos Longevity Research Institute
Other Study IDs: AG0119; 1R03AG030551-01A1 (NIH)
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Oxidative Stress; Aging
Keywords: VO2 max; stress; cortisol; fitness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fit
- Unfit

SUMMARY:
The purpose of this study is to test the hypothesis that physiological adaptations to regular exercise training (i.e. physical fitness) attenuates age-related decline in stress resilience to both oxidative stress and the neuroendocrine responses to psychosocial stress.

DETAILED DESCRIPTION:
Aging is associated with diminished stress resilience, as in reduced ability to manage or recover from acute changes in homeostasis. Increased oxidative damage to cells and tissues and dysregulation of stress hormones have been linked to age-associated chronic diseases including atherosclerosis, cancer, cardiovascular disease and Alzheimer's disease. Interventions to improve the body's resistance to stress, resulting in lower oxidative stress and better regulation of the stress hormones, may prevent or delay the onset of age-related diseases and improve quality of life.

Oxidative stress is believed to be a key mechanism in the aging process, with free radicals also implicated in many pathological processes. Similarly, dysregulation of the hypothalamic-pituitary-adrenal (HPA) axis is thought to play a role in aging and is linked to the increased risk for age-related chronic disease.

The hormesis theory suggests that a certain amount of stress can lead to better survival and reduced tissue damage following a subsequent, more severe stress. One way to stress the system is through acute exercise. Regular exercise training, however, results in adaptive responses that increase the tolerance for successive (exercise) stress.

A relevant question is whether adaptations to regular exercise training translate to greater resilience to psychosocial stress and an increased capacity to resist acute oxidative stress, thereby providing increased protection from diseases associated with dysregulation of these systems.

This study will investigate stress resilience in two areas related to aging: oxidative stress and the neuroendocrine response to psychosocial stress. The effects of physical fitness on oxidative stress compensation and neuroendocrine stress reactivity will be determined by comparing fit and unfit older men and women. The overall aim of this study is to provide enhanced understanding of the mechanisms by which physical fitness modifies stress resilience in older men and women.

ELIGIBILITY:
Inclusion Criteria:

* Men and post-menopausal women, ages 60-80 years
* Generally good health by self-report

Exclusion Criteria:

* Estrogen or testosterone supplementation within the previous 6 months
* Current smoker
* Body Mass Index (BMI) > 32 kg/m2
* Any chronic illness that could affect cortisol levels, including diabetes mellitus, liver or renal disease
* Evidence of a previous myocardial infarction within the last 6 months by EKG or history of angina or shortness of breath
* Clinically significant arrhythmia on a resting EKG or significant EKG changes during the baseline VO2max test
* Any other condition that would contraindicate maximal exercise testing, including elevated blood pressure at rest (systolic BP >140 or diastolic BP >90 mm Hg on at least 2 measurements, at least 10 minutes apart) or musculoskeletal problems
* Depression as measured by the Beck Depression Inventory (BDI score >17)
* Use of anti-oxidant supplements, in excess of standard multi-vitamins (1 tablet/day)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
F2-isoprostane response to an oxidative challenge (forearm ischemia-reperfusion trial) | Visit 4
Cortisol response (plasma and salivary) to a psychosocial laboratory stressor--Trier Social Stress Test (TSST) | Visit 3

SECONDARY OUTCOMES:
Total antioxidant capacity | Visit 4
ACTH response to TSST | Visit 3
Heart rate response to the TSST | Visit 3

CONTACTS AND LOCATIONS:
Overall Officials: Tinna Traustadóttir, PhD, Principal Investigator — Kronos Longevity Research Institute
Locations (1):
- Kronos Longevity Research Institute, Phoenix, Arizona, United States

REFERENCES:
- [Background] Traustadottir T, Bosch PR, Matt KS. The HPA axis response to stress in women: effects of aging and fitness. Psychoneuroendocrinology. 2005 May;30(4):392-402. doi: 10.1016/j.psyneuen.2004.11.002. Epub 2005 Jan 11. PMID 15694119
- [Background] Fatouros IG, Jamurtas AZ, Villiotou V, Pouliopoulou S, Fotinakis P, Taxildaris K, Deliconstantinos G. Oxidative stress responses in older men during endurance training and detraining. Med Sci Sports Exerc. 2004 Dec;36(12):2065-72. doi: 10.1249/01.mss.0000147632.17450.ff. PMID 15570141
- [Background] Vincent HK, Bourguignon C, Vincent KR. Resistance training lowers exercise-induced oxidative stress and homocysteine levels in overweight and obese older adults. Obesity (Silver Spring). 2006 Nov;14(11):1921-30. doi: 10.1038/oby.2006.224. PMID 17135607
- [Background] Finkel T, Holbrook NJ. Oxidants, oxidative stress and the biology of ageing. Nature. 2000 Nov 9;408(6809):239-47. doi: 10.1038/35041687. PMID 11089981
- See also: Kronos Longevity Research Institute — http://www.kronosinstitute.org